CLINICAL TRIAL: NCT00000398
Title: Behavioral Treatment of Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AR044064 (NIH); R01AR044064 (NIH); NIAMS-032
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2000-06

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Pain; Coping skills training; Physical exercise training; Combined coping skills training and exercise training
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Exercise

INTERVENTIONS:
Behavioral: Coping skills training
Behavioral: Physical exercise training
Behavioral: Coping skills training plus physical exercise training

SUMMARY:
Fibromyalgia (FM) is one of the most common rheumatic diseases (conditions or disorders that cause pain or stiffness in the joints, muscles, or bones). It affects 6 million Americans and up to 20 percent of patients seen by doctors who specialize in treating rheumatic diseases. This study will evaluate the effects of two of the most promising nondrug treatments for FM: coping skills training and physical exercise training. We will randomly assign each of 180 patients diagnosed with FM to one of four groups: coping skills training (CST), physical exercise training alone, CST plus physical exercise training, or a waiting list (nontreatment group). We will look at the separate and combined effects of CST and physical exercise training and evaluate how changes in aerobic fitness, self-effectiveness (a person's belief in his or her ability to reach a goal, such as managing one's own disease), and negative pain-related thoughts relate to improvements in pain and disability.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is characterized by diffuse musculoskeletal pain, discrete tender points at typical soft-tissue sites, fatigue, stiffness, and sleep problems. Of these symptoms, pain is often the primary concern of FM patients and their physicians. Traditional medical approaches to managing FM have limitations (side effects) and have not been effective in managing pain. Given these limitations, treatments that involve nonpharmacologic interventions may represent a valuable addition to patient care. This study will evaluate the effects of two of the most promising nonpharmacologic interventions for FM: coping skills training (CST) for pain management and physical exercise training.

The study is designed to test the hypothesis that an intervention that combines CST and physical exercise training will be more effective than CST or exercise alone. In this study, we will randomly assign each of 180 patients diagnosed with FM to one of four conditions: CST alone, physical exercise training alone, CST plus physical exercise training, or a waiting list control. We will evaluate study participants on four occasions: pre-treatment, post-treatment, 3-month followup, and 6-month followup.

The study will look at the separate and combined effects of CST and physical exercise training and evaluate how changes in aerobic fitness, self-effectiveness, and negative pain-related thoughts relate to improvements in pain and disability. Physicians could use this information in matching FM patients to treatment interventions. In addition, our findings may have implications for treatment selection for a broad range of patients suffering from persistent pain.

ELIGIBILITY:
Inclusion Criteria:

* Complaints of pain persisting for 6 months
* Meet diagnostic criteria for fibromyalgia (American College of Rheumatology criteria)

Exclusion Criteria:

* A significant adverse medical condition that would expose the individual to increased risk of an adverse experience during the course of the trial (e.g. a recent (<6 months) myocardial infarction)
* An abnormal cardiac response to exercise
* Other significant rheumatic disease
* Receiving or applying for disability or compensation benefits because of fibromyalgia

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 1996-07; Study Completion 2000-06

CONTACTS AND LOCATIONS:
Overall Officials: Christopher France, PhD, Principal Investigator — Ohio University
Locations (2):
- United States (2):
  - Ohio University, Athens, Ohio
  - Ohio State University, Columbus, Ohio

REFERENCES:
- [Background] Lester, N., and F.J. Keefe. "Coping With Chronic Pain." In Cambridge Handbook of Psychology, Health and Medicine, edited by A. Baum, C. McManus, S. Newman, J. Weinman, and R. West. Cambridge, England: Cambridge University Press, 1997.
- [Background] Sandstrom MJ, Keefe FJ. Self-management of fibromyalgia: the role of formal coping skills training and physical exercise training programs. Arthritis Care Res. 1998 Dec;11(6):432-47. doi: 10.1002/art.1790110603. PMID 10030175
- [Background] Keefe, F.J., France, C. Pain: Biopsychosocial mechanisms and management. Current Directions in Psychological Science 1999; 8:137-141.
- [Background] Keefe FJ, Bonk V. Psychosocial assessment of pain in patients having rheumatic diseases. Rheum Dis Clin North Am. 1999 Feb;25(1):81-103. doi: 10.1016/s0889-857x(05)70056-9. PMID 10083960
- [Background] Keefe FJ, Jacobs M, Underwood-Gordon L. Biobehavioral pain research: a multi-institute assessment of cross-cutting issues and research needs. Clin J Pain. 1997 Jun;13(2):91-103. doi: 10.1097/00002508-199706000-00003. PMID 9186016
- [Background] Keefe, F.J. "Cognitive Processes and the Pain Experience." In Journal of Musculoskeletal Pain, edited by S.R. Pillemer. 1998; 6:41-45.